CLINICAL TRIAL: NCT03097692
Title: Variable Types of Preconditioning,is There a Different Impact Upon Multiorgan Function After Open Heart Surgery ?
Brief Title: Does Preconditioning Affects Other Organs in Patients Undergoing Open Heart Surgery ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00009909
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Neutrophil Lymphocyte Ratio; Serum Createnine; Mechanical Ventilation
Keywords: cardiac preconditioning; open heart surgery; createnine; inflammation
MeSH Terms: conditions — Inflammation | interventions — Ischemic Preconditioning

STUDY DESIGN:
Intervention Model Description: intervention group well be pretreated with cardiac preconditioning
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic preconditioing (Active Comparator): 50 patients ischemic preconditioning will be done after induction and before cardiopulmonary bypass by inflation the cuff of blood pressure above 200mmhg in the lower limb every 5 min for 3cycles
  Interventions: Procedure: ischemic preconditioning
- Pharmacologic preconditioing (Active Comparator): by sevoflurane anesthesia
  Interventions: Drug: Pharmacologic preconditionig

INTERVENTIONS:
Procedure: ischemic preconditioning — ischemic preconditioning will be done after induction and before cardiopulmonary bypass by inflation the cuff of blood pressure above 200mmhg in the lower limb every 5 min for 3cycles
  Arms: Ischemic preconditioing
Drug: Pharmacologic preconditionig — Pharmacologic preconditionig will be attained by sevoflurane anesthesia
  Arms: Pharmacologic preconditioing

SUMMARY:
An association between white blood cell count (WBC), neutrophil-lymphocyte ratio , and inflammatory process is well known . Ischemic preconditioning reduces the inflammation

DETAILED DESCRIPTION:
Preliminary evidence has suggested the role of inflammation in development and prognosis of cardiovascular diseases and cancers. Most of the prognostic studies failed to account for the effects of co-morbid conditions as these might have raised the systemic inflammation. We used neutrophil lymphocyte ratio (NLR) as a measure of systemic inflammation and investigated its association with cardiac preconditioning in open heart surgery .

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* American Society of Anesthesiologists physical status II and III
* Patients scheduled for open heart surgery
* no active inflammatory process

Exclusion Criteria:Exclusion Criteria:

* Emergency surgery
* Clinically significant kidney or liver disease
* Patients allergic to local anesthetic
* Patients with prolonged cardiopulmonary bypass time (>120 min)
* Patients required intra-aortic balloon pump
* Postoperative hemodynamic instability (including the occurrence of serious arrhythmia) or bleeding that required surgical re-exploration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
change of Neutrophil lymphocyte ratio | during first two postoperative days

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided